CLINICAL TRIAL: NCT03235700
Title: Hyperemic Efficacy of Intravenous Infusion of Adenosine in Heart Failure With Reduced Ejection Fraction
Brief Title: Hyperemic Efficacy of IV Adenosine in HFrEF
Acronym: HF-FFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sejong General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1642
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Coronary Artery Disease
Keywords: heart failure with reduced ejection fraction; intermediate coronary stenosis; adenosine; hyperemia
MeSH Terms: conditions — Coronary Artery Disease; Hyperemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adenosine followed by nicorandil (Experimental)
  Interventions: Other: Maximal hyperemia with adenosine followed by nicorandil
- Nicorandil followed by adenosine (Experimental)
  Interventions: Other: Maximal hyperemia with nicorandil followed by adenosine

INTERVENTIONS:
Other: Maximal hyperemia with adenosine followed by nicorandil — IV adenosine 140 - IV adenosine 180 - IC adenosine (LCA 200/RCA 100) - IC nicorandil 2
  Arms: Adenosine followed by nicorandil
Other: Maximal hyperemia with nicorandil followed by adenosine — IC nicorandil 2 - IV adenosine 140 - IV adenosine 180 - IC adenosine (LCA 200/RCA 100)
  Arms: Nicorandil followed by adenosine

SUMMARY:
Little is known about the hyperemic efficacy of IV adenosine as well as safety in patients with heart failure with reduced ejection fraction (HFrEF) because they were excluded from the major FFR studies. We will evaluate the feasibility and hyperemic efficacy of IV adenosine in patients with HFrEF in comparison with IC nicorandil for invasive physiological assessment using a coronary pressure wire.

DETAILED DESCRIPTION:
Little is known about the hyperemic efficacy of IV adenosine as well as safety in patients with heart failure with reduced ejection fraction (HFrEF) because they were excluded from the major FFR studies. We will evaluate the feasibility and hyperemic efficacy of IV adenosine in patients with HFrEF in comparison with IC nicorandil for invasive physiological assessment using a coronary pressure wire. Patients with an angiographically intermediate lesion (40-70% diameter stenosis) in a major epicardial coronary artery and with left ventricle ejection fraction ≤40% will be prospectively enrolled. FFR under the various hyperemic stimulation using IV adenosine 140 & 180, IC adenosine, and IC nicorandil will be measured sequentially.

ELIGIBILITY:
Inclusion Criteria:

* angiographically proven epicardial intermediate stenosis (40-70%)
* echocardiographically proven LV dysfunction (LVEF ≤40%)

Exclusion Criteria:

* infarct-related artery, less than 2 weeks
* Killip class 3 and 4
* bronchial asthma
* second degree or third degree AV block
* any contraindications to adenosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Failure to induce maximal hyperemia | less than 1 day
  no hyperemia, cyclic hyperemia, and submaximal hyperemia

SECONDARY OUTCOMES:
Fractional flow reserve | less than 1 day
time to maximal hyperemia | less than 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Sejong general hospital, 91-121 Sosa 2-Dong, Sosa-Gu, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided